CLINICAL TRIAL: NCT03371641
Title: In Utero Alcoholic Exposure: PlGF, Biomarker of Fetal Brain Lesions
Acronym: ALCOBRAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016/0337/HP
Record Dates: First submitted 2017-11-29; First posted 2017-12-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Fetal Alcohol Syndrome
Keywords: Fetal Alcohol Syndrome; Pregnancy; Biomarker; PlGF; Cognitive development; Behavior troubles
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcoholic exposure group (Other): Blood sample (mother) Cord blood sample Placenta sample ASQ parental questionnaire WPPSI - IV and NEPSY development scales Scale of Conners SCQ questionnaire
  Interventions: Behavioral: ASQ parental questionnaire; Behavioral: Development scales; Behavioral: Scale of Conners; Behavioral: SCQ Questionnaire; Procedure: Blood sample (mother); Procedure: Cord blood sample; Procedure: Placenta sample
- Control (Other): Blood sample (mother) Cord blood sample Placenta sample ASQ parental questionnaire WPPSI - IV and NEPSY development scales Scale of Conners SCQ questionnaire
  Interventions: Behavioral: ASQ parental questionnaire; Behavioral: Development scales; Behavioral: Scale of Conners; Behavioral: SCQ Questionnaire; Procedure: Blood sample (mother); Procedure: Cord blood sample; Procedure: Placenta sample

INTERVENTIONS:
Behavioral: ASQ parental questionnaire — ASQ parental questionnaire
Behavioral: Development scales — WPPSI - IV and NEPSY development scales
Behavioral: Scale of Conners — Scale of Conners
Behavioral: SCQ Questionnaire — SCQ questionnaire
Procedure: Blood sample (mother) — Blood sample (mother) before delivery
Procedure: Cord blood sample — Cord blood sample after delivery
Procedure: Placenta sample — Placenta sample

SUMMARY:
This study aims to validate that PLGF is a biomarker of cerebral lesions and therefore of secondary developmental disorders and disabilities that will be best diagnosed at 2 and 6 years of age.

ELIGIBILITY:
Inclusion Criteria:

Mother:

* Pregnant woman (monofetal or twin pregnancy, whatever the parity)
* Age> or = to 18 years
* Person affiliated to a social security system
* Person who read and understood the information form and signed the consent form

  * Alcohol exposure group Chronic consumption of at least 30 g of alcohol per week or acute consumption of "binge drinking" type during pregnancy (knowing that a unit of 10 g of pure alcohol corresponds to 25 cl of beer 4 ° 5, 10 cl of wine at 12 °, 3 cl of whiskey, 7 cl of Porto ...)
  * Control group No alcohol consumption during pregnancy
  * Child Informed parents and written consent signed by the father and mother for the child's participation in this research (unless one of the parents does not have parental authority)

Exclusion Criteria:

* Female under 18
* Pregnant woman with clinical suspicion of pre-eclampsia and / or HELLP syndrome
* Person deprived of liberty by an administrative or judicial decision or protected major subject (under tutorship or curatorship)
* Patient participating in another interventional trial or who participated in another interventional trial during pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01-27 (Actual); Primary Completion 2026-03-27 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
PLGF concentrations in the umbilical cord | Through inclusion completion and samples analyses, an average of 4 months after the end of inclusions
  Compare concentrations between 2 groups of mother / child pairs: in utero exposure to alcohol versus control.
PLGF concentrations in placenta | Through inclusion completion and samples analyses, an average of 4 months after the end of inclusions
  Compare concentrations between 2 groups of mother / child pairs: in utero exposure to alcohol versus control.

SECONDARY OUTCOMES:
Assessment of the concentration of PLGF in maternal blood | Through inclusion completion and samples analyses, an average of 4 months after the end of inclusions
  Blood sample
Studies of metabolomic profile on blood sample | Through inclusion completion and samples analyses, an average of 4 months after the end of inclusions
  blood sample metabolomic profile
Studies of metabolomic profile on placenta | Through inclusion completion and samples analyses, an average of 4 months after the end of inclusions
  placenta metabolomic profile
Neurological clinical evaluation | The day of birth
  Clinical exam
Follow-up at 2 years in pediatric consultation for evaluation of neuro-development | 2 years
  ASQ: Ages & Stages Questionnaires. This questionnaire screens and assesses the developmental performance of children in the areas of communication, gross motor skills, fine motor skills, problem solving, and personal-social skills. It is used to identify children that would benefit from in-depth evaluation for developmental delays.
Follow-up at 6 years in consultation for assessment of neurodevelopment with | 6 years
  parental ASQ: Ages & Stages Questionnaire screens and assesses the developmental performance of children in the areas of communication, gross motor skills, fine motor skills, problem solving, and personal-social skills. It is used to identify children that would benefit from in-depth evaluation for developmental delays.
Follow-up at 6 years in consultation for assessment of neuropsychological assessment: Wechsler Preschool and Primary Scale of Intelligence: WPPSI IV | 6 years
  WPPSI - IV: The Wechsler Preschool and Primary Scale of Intelligence consist of 14 subtests. They are designated as one of three types: core, supplemental, or optional. The core subtests are required for the computation of the Verbal, Performance, and Full Scale IQ. The supplemental subtests provide additional information about cognitive abilities or can be used as replacement for inappropriate subtests. The optional subtests provide additional information about cognitive functioning but cannot be used as replacements for core subtests. Quotient and Composite scores have a mean of 100 and a standard deviation of 15. Subtest scaled scores have a mean of 10 and a standard deviation of 3.elow 70 is Extremely Low, 70-79 is Borderline, 80-89 is Low Average, 90-109 is Average, 110-119 is High Average, 120-129 is Superior, 130+ is Very Superior.
Follow-up at 6 years in consultation for assessment of neuropsychological assessment: Developmental NEuroPSYchological Assessment | 6 years
  NEPSY -NEuroPSYchological Assessment. The six functional domains are made up of 32 subtests and four delayed tasks. These domains are theoretically, not statistically, derived. The subtests were designed to assess cognitive abilities related to disorders that are typically diagnosed in childhood and that are required for success in an academic environment. These tests supposedly help detect any underlying deficiencies that may impede a child's learning
Follow-up at 6 years in consultation for assessment of neuropsychological assessment: Conners' scale | 6 years
  Conners scale is assessing for attention deficit hyperactivity disorder (ADHD)
Follow-up at 6 years in consultation for assessment of neuropsychological assessment: SCQ Social Communication Questionnaire | 6 years
  SCQ: The Social Communication is a 40 item, parent report screening measure that taps the symptomatology associaed with autism Spectrum disorder (ASD). The items are administered in a yes/non response format.

CONTACTS AND LOCATIONS:
Locations (1):
- UH ROUEN, Rouen, France

IPD SHARING:
Plan to Share IPD: No